CLINICAL TRIAL: NCT03892759
Title: Osteopathic Manipulative Treatment for Back Pain: Evaluation of Short Term Changes in Functional Status, Quality of Life, and Pain
Brief Title: Osteopathic Manipulative Treatment for Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Northwest University of Health Sciences (Other)
Responsible Party: Principal Investigator, Crystal Martin, Principal Investigator, Pacific Northwest University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-006
Record Dates: First submitted 2019-03-22; First posted 2019-03-27 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Back Pain; Lumbar Pain; Thoracic Pain; Somatic Dysfunction; Fascial Distortion
Keywords: Osteopathic Manipulative Treatment
MeSH Terms: conditions — Back Pain; Low Back Pain; Chest Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Pre/post prospective one group pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation and Treatment (Other): Subjects will be evaluated through inspection and palpation of the thoracic and lumbar spine, and other body regions as necessary. The provider will make a diagnosis of somatic dysfunction based off the TART (tissue texture change, asymmetry, restriction of motion, tenderness/pain) findings.
  Interventions: Other: Osteopathic Manipulative Therapy

INTERVENTIONS:
Other: Osteopathic Manipulative Therapy — A set of hands-on techniques used by Osteopathic Physicians for the assessment and treatment of somatic dysfunction.

SUMMARY:
This study will investigate if Osteopathic Manipulative Treatment (OMT) is beneficial for patients presenting with back pain.

DETAILED DESCRIPTION:
Low back pain is the most common cause of disability in people under age 45 and accounts for 20% of all physician visits. Osteopathic manual treatment (OMT) has been used to manage patients with acute and chronic back pain. These treatments are often reported as beneficial by patients.

This study will examine the effect on functional status, range of motion, quality of life, and pain with Osteopathic Manipulative Treatment (OMT). Baseline will be defined as someone who has never had OMT, chiropractic, or massage, or has not received such treatments in the last 90 days. Back pain will be specific to pain presenting in the lumbar or thoracic regions of the spine.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older
* Back pain
* Able to arrange transportation and arrive to three study appointments.

Exclusion Criteria:

* May not have had manual treatment (massage, chiropractic, or OMT) in the last 90 days
* May not have any labs or imaging for their back pain recommended by their physicians the subject has not yet completed
* May not have had back surgery in past 60 days
* May not be pregnant or have given birth in the last 30 days
* May not have be unable to tell a member of the study team their name, city they live in and the current year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Functional Status at 8 weeks | 8 weeks
  Functional Status as measured by Roland-Morris Disability Questionnaire. Question responses are totaled for a score of 0 to 24 with higher number indicating a worse outcome or greater level of disability.
Change from Baseline Functional Status at 12 weeks | 12 weeks
  Functional Status as measured by Roland-Morris Disability Questionnaire. Question responses are totaled for a score of 0 to 24 with higher number indicating a worse outcome or greater level of disability.
Change from Baseline Back Range of Motion at 3 weeks | 3 Weeks
  Range of Motion a measured by Back Range of Motion (BROM) Instrument
Change from Baseline Back Range of Motion at 8 weeks | 8 weeks
  Range of Motion a measured by Back Range of Motion (BROM) Instrument
Change from Baseline Back Pain at 3 weeks | 3 weeks
  Pain as measured by Visual Analog Scale (VAS). The scale indicates a level of pain from 0 to 10 with higher number associated with a worse outcome or greater level of pain.
Change from Baseline Back Pain at 8 weeks | 8 weeks
  Pain as measured by Visual Analog Scale (VAS). The scale indicates a level of pain from 0 to 10 with higher number associated with a worse outcome or greater level of pain.

SECONDARY OUTCOMES:
Change from Baseline Assessment of Quality of Life at 8 weeks | 8 weeks
  Quality of Life as measured by PROMIS Global Health Questionnaire. Total Physical Health Score of 7 to 17 with lower numbers indicating better physical health outcome and Total Mental Health Score of 8 to 16 with lower numbers indicating better mental health outcome.
Change from Baseline Assessment of Quality of Life at 12 weeks | 12 weeks
  Quality of Life as measured by PROMIS Global Health Questionnaire. Total Physical Health Score of 7 to 17 with lower numbers indicating better physical health outcome and Total Mental Health Score of 8 to 16 with lower numbers indicating better mental health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Martin, DO, Principal Investigator — Assistant Professor of Osteopathic Principles and Practice
Locations (1):
- Pacific Northwest University of Health Sciences, Yakima, Washington, United States